CLINICAL TRIAL: NCT02860494
Title: Topical Everolimus Versus Placebo for the Treatment of Facial Angiofibromas in Patients With Tuberous Sclerosis Complex. A Phase II/III, Multicentre, Randomized, Double-blind, Placebo-controlled Study of 3 Doses of Topical Everolimus.
Brief Title: Topical Everolimus in Patients With Tuberous Sclerosis Complex
Acronym: EVEROST
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Pharmaceutical and financial difficulties
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL16_0062; 2018-002531-18 (EudraCT Number)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Facial Angiofibromas
Keywords: Tuberous sclerosis complex (TSC); topical everolimus; seamless design; dose-escalation study; m-TOR inhibitor
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Topical everolimus 0.1% (Experimental): Everolimus topical formulation will be applied to the affected areas, once daily, in the evening, for 6 months. Dose regimens will be identical, regardless of the dose-strength of the topical formulation. The topical formulation will be applied onto areas of the face affected by FA by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Interventions: Drug: Everolimus
- Topical everolimus 0.5% (Experimental): Everolimus topical formulation will be applied to the affected areas, once daily, in the evening, for 6 months. Dose regimens will be identical, regardless of the dose-strength of the topical formulation. The topical formulation will be applied onto areas of the face affected by FA by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Interventions: Drug: Everolimus
- Topical everolimus 1% (Experimental): Everolimus topical formulation will be applied to the affected areas, once daily, in the evening, for 6 months. Dose regimens will be identical, regardless of the dose-strength of the topical formulation. The topical formulation will be applied onto areas of the face affected by FA by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Interventions: Drug: Everolimus
- Topical placebo (Placebo Comparator): Topical placebo will be identical to the everolimus topical formulation. Topical placebo will be applied to the affected areas, once daily, in the evening, for 6 months by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus topical formulation will be applied to the affected areas, once daily, in the evening, for 6 months. Dose regimens will be identical, regardless of the dose-strength of the topical formulation. The topical formulation will be applied onto areas of the face affected by FA by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Arms: Topical everolimus 0.1%; Topical everolimus 0.5%; Topical everolimus 1%
Drug: Placebo — Placebo topical formulation will be applied to the affected areas, once daily, in the evening, for 6 months, by the patient or the patient's parents/legal guardians, while observing standardised precautions (avoiding the eyes, washing the hands after application, etc.).
  Arms: Topical placebo

SUMMARY:
Tuberous sclerosis complex (TSC) is a rare genetic multisystem disorder characterized by the development of hamartomas in several organs (e.g. brain, heart, kidney, liver, lung), and skin in more than 90% of cases. Facial angiofibromas (FA), present in about 80% of patients, are a stigmatizing hallmark of the disease. Everolimus could be a candidate for use as a topical formulation to treat FA. This adaptive seamless Phase II/III study primary objective is to determine the dose of topical everolimus for treatment of FA and evaluate the efficacy and safety of topical everolimus versus placebo in patients with angiofibromas.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 2 years
* With definite or possible diagnosis of TSC
* With at least 3 FA, diagnosed by a dermatologist
* Patients (or parents or legal guardians) who have provided written informed consent prior to participation in the study
* Willing and able to comply with study requirements
* With negative blood pregnancy test at the screening visit and using effective contraceptive methods for women of childbearing potential, up to 12 weeks after treatment discontinuation
* Covered by national health insurance

Exclusion Criteria:

* Systemic treatment by sirolimus, everolimus, or any other immunosuppressive drug, during the previous 6 months
* Use of topical tacrolimus or sirolimus on the face, during the previous 6 months
* Destructive treatment (laser therapy, surgery, cryotherapy) of facial angiofibromas during the previous 6 months
* Concomitant use of topical treatments that could affect facial erythema (e.g. Brimonidine)
* Known internal organ involvement requiring systemic mTOR inhibitor in the next 6 months
* Immunosuppression (immunosuppressive disease or immunosuppressive treatment)
* Known chronic infectious disease Known hypersensitivity to mTOR inhibitor
* Neutropenia < 1000/mm3
* Thrombopenia < 75,000/mm3
* Chronic renal insufficiency (estimated Glomerular Filtration Rate < 60 mls/min)
* Chronic liver disease (SGOT or SGPT > 3 times upper normal limit)
* Uncontrolled dyslipidaemia
* Uncontrolled diabetes
* Brest feeding or pregnant women, or women on childbearing age without any effective method of contraception during treatment and up to 12 weeks after treatment discontinuation
* Subjects who, in the Investigator's opinion, are unable or unwilling to comply with the protocol.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Facial Angiofibroma Severity Index (FASI) | 6 months
  The FASI is a composite score summing the scores for erythema (0-3), size (0-3) and extension of FA (2:<50% of the cheek surface; 3:>50% of the cheek surface). The FASI will be centrally-measured on patient's face photographs by an independent and blinded adjudication committee of 2 dermatologists, with third-dermatologist review for disagreements.

SECONDARY OUTCOMES:
FA size | 6 months
  FA size (in millimetres) of the 3 largest targeted FA papules previously identified by the investigator
Dermatologist's global assessment of efficacy | 6 months
  using 7-point Likert scale
Patient or parents self-assessment | 6 months
  using 7-point Likert scale
Local tolerance of the topically applied formulation using patient self-assessment | 6 months
blood levels of topically applied everolimus | 6 months
dryness score | 6 months
  assessed by physicians
scaling scores | 6 months
  assessed by physicians
Dermatological quality of life | 6 months
  using DLQI (Dermatology Life Quality Index) for adults, CDLQI (Children's Dermatology Life Quality Index) for children

CONTACTS AND LOCATIONS:
Overall Officials: Alice PHAN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No